CLINICAL TRIAL: NCT03733639
Title: The Use of Fibrin Glue Sealant (Tisseel®) as a Reinforcement of Esophagojejunal Anastomoses Will Decrease the Rate of Anastomotic Leak.
Brief Title: Tisseel® as a Reinforcement of Esophagojejunal Anastomoses
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Germans Trias i Pujol Hospital (Other)
Responsible Party: Principal Investigator, Elisenda Garsot Savall, Head of Upper Gastrointestinal Surgery Unit, Germans Trias i Pujol Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Tisseel
Record Dates: First submitted 2018-10-18; First posted 2018-11-07 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Gastric Cancer; Anastomotic Leak
MeSH Terms: conditions — Stomach Neoplasms; Anastomotic Leak | interventions — Fibrin Tissue Adhesive

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients won't know if his anastomoses has been reinforced with Tisseel®.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Tisseel® (Active Comparator): Once the esophagojejunal anastomosis is done the patient is randomized (Tisseel® vs no product). In the arm "Tisseel®" surgeon dispenses the product all over the anastomosis. The rest of the surgical procedure is as usual.
  Interventions: Drug: Tisseel
- no Tisseel® (Other): Once the esophagojejunal anastomosis is done the patient is randomized (Tisseel® vs no product). In the arm " noTisseel®" surgeon performs the surgical procedure as usual.
  Interventions: Device: No Tisseel

INTERVENTIONS:
Drug: Tisseel — Reinforcement of esophagojejunal anastomoses after total gastrectomy with the product.
  Arms: Tisseel®
Device: No Tisseel — No reinforcement of esophagojejunal anastomoses after total gastrectomy
  Arms: no Tisseel®

SUMMARY:
Background:

The dehiscence of esophagojejunal anastomoses is one of the most serious complications after total gastrectomy in patients with gastric cancer. Any method of avoiding this problem will affect not only the postoperative course but also the prognostic of disease.

Methods:

This is a prospective, randomized and multicenter trial, within the Spanish EURECCA Esophagogastric Cancer Group, to investigate the efficacy of Tisseel® in reducing the rate of esophagojejunal anastomosis leakage in patients with gastric cancer. The rate of anastomosis leak will be measured with clinical, radiological and analytic parameters.

Objective:

Analyze the efficacy of Tisseel® as a reinforcement in reducing the rate of anastomotic esophagojejunal anastomoses.

DETAILED DESCRIPTION:
Introduction The dehiscence of the esophagojejunal anastomosis is one of the most serious complications after a total gastrectomy not only in the short term but it has been shown to be an independent risk factor for survival. The rate of esophagojejunal anastomosis leakage after cancer gastrectomies is described to be between 1-12.3%.

Any method to prevent this complication would be of vital importance to improve the evolution of these patients. Likewise, when the dehiscence has been established, early detection could contribute to an early intervention, avoiding more serious consequences and, therefore, improving the short and long term prognosis.

Little progress has been made during recent decades in the prevention of anastomotic leakage in high-risk digestive tract anastomosis. Some authors have tried the use of new methods of suture, reinforcements or patches in the anastomosis. Fibrin adhesives were introduced more than 30 years ago, in order to favor hemostasis and tissue adhesion. Numerous studies have demonstrated their effectiveness in reducing surgical bleeding in cardiovascular surgery but its role as a sealant in gastrointestinal anastomosis is more debated. There have been some experimental studies that have shown a possible protective effect of this material in enteric anastomoses. With the evolution of bariatric surgery and with the high volume of surgeries handled, several studies have been published that assess the effect of fibrin sealants on gastrojejunal anastomoses. In esophagogastric surgery, the number of published studies is reduced and there are only 2 studies that assess the effect of fibrin sealants on esophagojejunal anastomosis. The results of these studies seem to indicate that the application of fibrin sealants in this anastomosis could have a favorable effect in reducing the number of anastomotic dehiscences.

There are different definitions for the concept of "anastomotic dehiscence". The dehiscence of the esophago-jejunal anastomotic can be defined as any clinical and / or radiological evidence of dehiscence of the anastomosis. Although early diagnosis is key to avoiding major consequences, in clinical practice, the diagnosis of anastomotic dehiscence is often delayed. Direct observation of the debit of surgical drainage, fever or persistent ileus or clear symptoms of peritonitis are indirect signs that make us suspect a possible anastomotic dehiscence. The possibility of having a parameter that allows us to diagnose early a problem in the suture would allow us to act earlier and, therefore, improve the prognosis of these patients in the short and long term.

In colorectal surgery, serological parameters such as procalcitonin or C-reactive protein have been studied as early predictors of anastomotic dehiscence. In esophagogastric surgery, publications are scarce and all of them analyze results in esophagogastric anastomoses.

Furthermore, the determination of amylases in drainage has also been used for the detection of postoperative fistula. It is a simple and low cost method and is a parameter widely used in pancreatic surgery for the detection and evolutionary control of pancreatic fistulas. It has also been shown to be useful in esophageal surgery and in bariatric surgery. However, in gastric cancer it has only been used for the diagnosis of pancreatic fistula as a complication in total gastrectomies with associated splenectomy.

Finally, the use of radiology with oral contrast routinely in the postoperative period of esophagogastric surgery has been shown to have a low sensitivity for the early detection of anastomotic dehiscence. CT with oral contrast seems to have greater sensitivity and positive predictive value in esophageal surgery for this purpose, but the need to perform a postoperative test to evaluate the anastomosis without clinical evidence of dehiscence is unclear.

For all these reasons, we believe that a multicenter randomized study will contribute to improve the clinical results of esophagogastric surgery and the knowledge of the diagnosis of complications, by studying the efficacy of Tisseel® in reducing the rate of anastomotic leakage, but also analyzing the role of drain amylases, serum CRP (C-reactive protein), procalcitonin and white blood cell levels in the early detection and prediction of anastomotic leak, and the role of CT with oral contrast as a routine assessment of anastomotic integrity.

Objective Analyze the efficacy of Tisseel® in reducing the rate of anastomotic leakage diagnosed in the postoperative period using clinical and / or radiological parameters.

Methods This is a prospective, randomized and multicenter trial, within the Spanish EURECCA Esophagogastric Cancer Project, to investigate the efficacy of Tisseel® in reducing the rate of esophagojejunal anastomosis leakage in patients with gastric cancer.

Participation study will be offered to all centers that are currently part of the Spanish EURECCA Esophagogastric Cancer Group. Those hospitals that show their desire to participate must sign the Letter of Commitment. In the same way, the study must sign off by European Medicine Agency and Spanish Agency of Medicines.

Once the patient is included in the study the surgeon performs a total gastrectomy as usual procedure. Once the esophagojejunal anastomosis is done the patient is randomized (Tisseel® vs no product). Surgeon dispenses Tisseel® all over the anastomosis following data sheet if applicable. The rest of the surgical procedure is as usual. In the postoperative period the investigator collects the data commented in following sections.

The evidence of an anastomotic leak will be tested with analytical and radiological parameters:

1. Blood samples will be taken from patients at:

   * Immediate preoperative (blood count, procalcitonin and C-reactive protein)
   * Days 1, 3, 5 and 7 postoperative (blood count, procalcitonin and C-reactive protein).
2. A sample of surgical drainage will be collected for the determination of amylases on days: 1,3,5, and 7 postoperative or until drainage is withdrawn.
3. An abdominal CT with oral contrast will be performed within the first 5 postoperative days. The date and the result will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years diagnosed with gastric adenocarcinoma and scheduled for a total gastrectomy with curative intent in EURECCA Esophagogastric Cancer Group who agree to participate in the study and sign the informed consent

Exclusion Criteria:

* Patients with non-epithelial neoplasms, with metastases, not resected or undergoing palliative resections. Patients who do not sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2020-07-21 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Rate of esophagojejunal anastomotic leak in immediate postoperative period | 7 days
  Clinical or radiological (see anex 1: Score Goense) evidence of esophagojejunal anastomotic leak.

SECONDARY OUTCOMES:
Amylases level in drainage | days 1,3,5,7 postoperatively
  Amylase level (mg/L) in drainage
CRP (C-reactive protein) in blood | days 1,3,5,7 postoperatively
  C-reactive protein in blood (mg/L)
Procalcitonin in blood | days 1,3,5,7 postoperatively
  Procalcitonin in blood (mg/L)
White cell levels in blood | days 1,3,5,7 postoperatively
  White cell levels in blood (x109/L)
Results of Computed Tomography with oral contrast. | between 3th and 5th postoperative day
  The results will be expressed based on Goense Score
  Based on Score Goense (Anastomotic Leakage Prediction Score). The investigator will collect the presence of:
  Yes No Normal Fluid collection Air cavity Fistula Wall discontinuity Empiema
  Goense L, Stassen PMC, Wessels FJ, van Rossum PSN, Ruurdal JP, van Leeuwen MS, van Hillegersberg R. Diagnostic performance of a CT-based scoring system for diagnosis of anastomotic leakage after esophagectomy: comparison with subjective CT assessment. Eur Radiol 2017; 27:4426-34
Type of esophagojejunal anastomoses performed | day of intervention
  The type of esophagojejunal anastomoses performed can be:
  1. mechanical (circular)
  2. mechanical (lineal)
  3. manual
Postoperative complications | 30 days after surgery
  Postoperative complications (Clavien-Dindo score):
  Grade I Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions
  Grade II Requiring pharmacological treatment with drugs other than such allowed for grade I complications.
  Grade III Requiring surgical, endoscopic or radiological intervention
  * IIIa Intervention not under general anesthesia
  * IIIb Intervention under general anesthesia
  Grade IV Life-threatening complication requiring IC/ICU-management
  * IVa single organ dysfunction (including dialysis)
  * IVb multiorgandysfunction
  Grade V Death of a patient
90-day mortality | 90 days after surgery
  Mortality at 90 days after surgery
Need for urgent surgical re-intervention | 30 days after surgery
  Reintervention after surgery:
  Yes/Not
Hospital stay | 30 days after surgery
  Number of days of hospital stay
Readmission | 30 days after discharge
  Readmission within 30 days after discharge:
  Yes/Not

CONTACTS AND LOCATIONS:
Overall Officials: Elisenda Garsot, Principal Investigator — Germans Trias i Pujol Hospital
Locations (1):
- Elisenda Garsot Savall, Badalona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aurello P, Magistri P, D'Angelo F, Valabrega S, Sirimarco D, Tierno SM, Nava AK, Ramacciato G. Treatment of esophagojejunal anastomosis leakage: a systematic review from the last two decades. Am Surg. 2015 May;81(5):450-3. PMID 25975326
- [Background] Migita K, Takayama T, Matsumoto S, Wakatsuki K, Enomoto K, Tanaka T, Ito M, Nakajima Y. Risk factors for esophagojejunal anastomotic leakage after elective gastrectomy for gastric cancer. J Gastrointest Surg. 2012 Sep;16(9):1659-65. doi: 10.1007/s11605-012-1932-4. Epub 2012 Jun 12. PMID 22688419
- [Background] De Stefano A, Bettarini F, Di Mare G, Neri A. [Enteric anastomosis and Tachosil(R)]. Minerva Chir. 2011 Jun;66(3):183-8. Italian. PMID 21666554
- [Background] Yuan Y, Zeng X, Hu Y, Xie T, Zhao Y. Omentoplasty for esophagogastrostomy after esophagectomy. Cochrane Database Syst Rev. 2012 Nov 14;11:CD008446. doi: 10.1002/14651858.CD008446.pub2. PMID 23152259
- [Background] Borst HG, Haverich A, Walterbusch G, Maatz W. Fibrin adhesive: an important hemostatic adjunct in cardiovascular operations. J Thorac Cardiovasc Surg. 1982 Oct;84(4):548-53. PMID 6981733
- [Background] Kjaergard HK, Fairbrother JE. Controlled clinical studies of fibrin sealant in cardiothoracic surgery--a review. Eur J Cardiothorac Surg. 1996;10(9):727-33. doi: 10.1016/s1010-7940(96)80332-0. PMID 8905274
- [Background] Matthew TL, Spotnitz WD, Kron IL, Daniel TM, Tribble CG, Nolan SP. Four years' experience with fibrin sealant in thoracic and cardiovascular surgery. Ann Thorac Surg. 1990 Jul;50(1):40-3; discussion 43-4. doi: 10.1016/0003-4975(90)90080-p. PMID 2369228
- [Background] Bonanomi G, Prince JM, McSteen F, Schauer PR, Hamad GG. Sealing effect of fibrin glue on the healing of gastrointestinal anastomoses: implications for the endoscopic treatment of leaks. Surg Endosc. 2004 Nov;18(11):1620-4. doi: 10.1007/s00464-004-8803-3. Epub 2004 Oct 11. PMID 15931477
- [Background] Silecchia G, Boru CE, Mouiel J, Rossi M, Anselmino M, Morino M, Toppino M, Gaspari A, Gentileschi P, Tacchino R, Basso N. The use of fibrin sealant to prevent major complications following laparoscopic gastric bypass: results of a multicenter, randomized trial. Surg Endosc. 2008 Nov;22(11):2492-7. doi: 10.1007/s00464-008-9885-0. Epub 2008 Mar 26. PMID 18365278
- [Background] Upadhyaya VD, Gopal SC, Gangopadhyaya AN, Gupta DK, Sharma S, Upadyaya A, Kumar V, Pandey A. Role of fibrin glue as a sealant to esophageal anastomosis in cases of congenital esophageal atresia with tracheoesophageal fistula. World J Surg. 2007 Dec;31(12):2412-5. doi: 10.1007/s00268-007-9244-7. PMID 17917772
- [Background] Saldana-Cortes JA, Larios-Arceo F, Prieto-Diaz-Chavez E, De Buen EP, Gonzalez-Mercado S, Alvarez-Villasenor AS, Prieto-Aldape MR, Fuentes-Orozco C, Gonzalez-Ojeda A. Role of fibrin glue in the prevention of cervical leakage and strictures after esophageal reconstruction of caustic injury. World J Surg. 2009 May;33(5):986-93. doi: 10.1007/s00268-009-9949-x. PMID 19234736
- [Background] Fernandez Fernandez L, Tejero E, Tieso A. Randomized trial of fibrin glue to seal mechanical oesophagojejunal anastomosis. Br J Surg. 1996 Jan;83(1):40-1. doi: 10.1002/bjs.1800830111. No abstract available. PMID 8653358
- [Background] Lago Oliver J, Arjona Medina I, Martin Garcia-Almenta E, Martin Gil J, Sanz Sanchez M, Perez Diaz MD, Alonso Poza A, Turegano Fuentes F, Torres Garcia A. [Use of fibrin based biological adhesives in the prevention of anastomotic leaks in the high risk digestive tract: preliminary results of the multicentre, prospective, randomised, controlled, and simple blind phase IV clinical trial: Protissucol001]. Cir Esp. 2012 Dec;90(10):647-55. doi: 10.1016/j.ciresp.2012.05.007. Epub 2012 Jun 27. Spanish. PMID 22748849
- [Background] Bruce J, Krukowski ZH, Al-Khairy G, Russell EM, Park KG. Systematic review of the definition and measurement of anastomotic leak after gastrointestinal surgery. Br J Surg. 2001 Sep;88(9):1157-68. doi: 10.1046/j.0007-1323.2001.01829.x. PMID 11531861
- [Background] Yoo HM, Lee HH, Shim JH, Jeon HM, Park CH, Song KY. Negative impact of leakage on survival of patients undergoing curative resection for advanced gastric cancer. J Surg Oncol. 2011 Dec;104(7):734-40. doi: 10.1002/jso.22045. Epub 2011 Jul 25. PMID 21792945
- [Background] Garcia-Granero A, Frasson M, Flor-Lorente B, Blanco F, Puga R, Carratala A, Garcia-Granero E. Procalcitonin and C-reactive protein as early predictors of anastomotic leak in colorectal surgery: a prospective observational study. Dis Colon Rectum. 2013 Apr;56(4):475-83. doi: 10.1097/DCR.0b013e31826ce825. PMID 23478615
- [Background] Giaccaglia V, Salvi PF, Antonelli MS, Nigri G, Pirozzi F, Casagranda B, Giacca M, Corcione F, de Manzini N, Balducci G, Ramacciato G. Procalcitonin Reveals Early Dehiscence in Colorectal Surgery: The PREDICS Study. Ann Surg. 2016 May;263(5):967-72. doi: 10.1097/SLA.0000000000001365. PMID 26528879
- [Background] Hayati F, Mohd Azman ZA, Nasuruddin DN, Mazlan L, Zakaria AD, Sagap I. Serum Procalcitonin Predicts Anastomotic Leaks in Colorectal Surgery. Asian Pac J Cancer Prev. 2017 Jul 27;18(7):1821-1825. doi: 10.22034/APJCP.2017.18.7.1821. PMID 28749112
- [Background] Noble F, Curtis N, Harris S, Kelly JJ, Bailey IS, Byrne JP, Underwood TJ; South Coast Cancer Collaboration-Oesophago-Gastric (SC-OG). Risk assessment using a novel score to predict anastomotic leak and major complications after oesophageal resection. J Gastrointest Surg. 2012 Jun;16(6):1083-95. doi: 10.1007/s11605-012-1867-9. Epub 2012 Mar 15. PMID 22419007
- [Background] Dutta S, Fullarton GM, Forshaw MJ, Horgan PG, McMillan DC. Persistent elevation of C-reactive protein following esophagogastric cancer resection as a predictor of postoperative surgical site infectious complications. World J Surg. 2011 May;35(5):1017-25. doi: 10.1007/s00268-011-1002-1. PMID 21350898
- [Background] Hoeboer SH, Groeneveld AB, Engels N, van Genderen M, Wijnhoven BP, van Bommel J. Rising C-reactive protein and procalcitonin levels precede early complications after esophagectomy. J Gastrointest Surg. 2015 Apr;19(4):613-24. doi: 10.1007/s11605-015-2745-z. Epub 2015 Feb 7. PMID 25663633
- [Background] Reid-Lombardo KM, Farnell MB, Crippa S, Barnett M, Maupin G, Bassi C, Traverso LW; Pancreatic Anastomotic Leak Study Group. Pancreatic anastomotic leakage after pancreaticoduodenectomy in 1,507 patients: a report from the Pancreatic Anastomotic Leak Study Group. J Gastrointest Surg. 2007 Nov;11(11):1451-8; discussion 1459. doi: 10.1007/s11605-007-0270-4. Epub 2007 Aug 21. PMID 17710506
- [Background] Perry Y, Towe CW, Kwong J, Ho VP, Linden PA. Serial Drain Amylase Can Accurately Detect Anastomotic Leak After Esophagectomy and May Facilitate Early Discharge. Ann Thorac Surg. 2015 Dec;100(6):2041-6; discussion 2046-7. doi: 10.1016/j.athoracsur.2015.05.092. Epub 2015 Aug 25. PMID 26319485
- [Background] Baker EH, Hill JS, Reames MK, Symanowski J, Hurley SC, Salo JC. Drain amylase aids detection of anastomotic leak after esophagectomy. J Gastrointest Oncol. 2016 Apr;7(2):181-8. doi: 10.3978/j.issn.2078-6891.2015.074. PMID 27034784
- [Background] Berkelmans GH, Kouwenhoven EA, Smeets BJ, Weijs TJ, Silva Corten LC, van Det MJ, Nieuwenhuijzen GA, Luyer MD. Diagnostic value of drain amylase for detecting intrathoracic leakage after esophagectomy. World J Gastroenterol. 2015 Aug 14;21(30):9118-25. doi: 10.3748/wjg.v21.i30.9118. PMID 26290638
- [Background] Maher JW, Bakhos W, Nahmias N, Wolfe LG, Meador JG, Baugh N, Kellum JM. Drain amylase levels are an adjunct in detection of gastrojejunostomy leaks after Roux-en-Y gastric bypass. J Am Coll Surg. 2009 May;208(5):881-4; discussion 885-6. doi: 10.1016/j.jamcollsurg.2008.12.022. Epub 2009 Mar 26. PMID 19476853
- [Background] Sano T, Sasako M, Katai H, Maruyama K. Amylase concentration of drainage fluid after total gastrectomy. Br J Surg. 1997 Sep;84(9):1310-2. PMID 9313722
- [Background] Cools-Lartigue J, Andalib A, Abo-Alsaud A, Gowing S, Nguyen M, Mulder D, Ferri L. Routine contrast esophagram has minimal impact on the postoperative management of patients undergoing esophagectomy for esophageal cancer. Ann Surg Oncol. 2014 Aug;21(8):2573-9. doi: 10.1245/s10434-014-3654-1. Epub 2014 Mar 28. PMID 24682648
- [Background] Struecker B, Chopra S, Heilmann AC, Spenke J, Denecke C, Sauer IM, Bahra M, Pratschke J, Andreou A, Biebl M. Routine Radiologic Contrast Agent Examination After Gastrectomy for Gastric Cancer Is Not Useful. J Gastrointest Surg. 2017 May;21(5):801-806. doi: 10.1007/s11605-017-3384-3. Epub 2017 Feb 15. PMID 28205124
- [Background] Strauss C, Mal F, Perniceni T, Bouzar N, Lenoir S, Gayet B, Palau R. Computed tomography versus water-soluble contrast swallow in the detection of intrathoracic anastomotic leak complicating esophagogastrectomy (Ivor Lewis): a prospective study in 97 patients. Ann Surg. 2010 Apr;251(4):647-51. doi: 10.1097/SLA.0b013e3181c1aeb8. PMID 19864934
- [Background] Jones CM, Clarke B, Heah R, Griffiths EA. Should routine assessment of anastomotic integrity be undertaken using radiological contrast swallow after oesophagectomy with intra-thoracic anastomosis? Best evidence topic (BET). Int J Surg. 2015 Aug;20:158-62. doi: 10.1016/j.ijsu.2015.06.076. Epub 2015 Jul 10. PMID 26166736